CLINICAL TRIAL: NCT02390102
Title: Combined ErythroPoietin and Iron Therapy for AnemiC Patients With Severe Symptomatic Aortic Stenosis Undergoing Transcatheter Aortic Valve REplacement- The EPICURE Trial A Prospective Double Blind Randomized Trial
Brief Title: Erythropoietin + Iron Therapy for Anemic Patients Undergoing Aortic Valve Replacement
Acronym: EPICURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, MD, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPICURE; CER-20809 (Other: Research Ethics Board)
Record Dates: First submitted 2013-01-21; First posted 2015-03-17 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Anemia; Aortic Stenosis
Keywords: Anemia; Severe aortic stenosis; Red blood cell transfusion; Erythropoietin
MeSH Terms: conditions — Anemia; Aortic Valve Stenosis | interventions — Erythropoietin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Erythropoietin (Active Comparator): Dose: darboepoetin 0.75µg/Kg + 200mg intravenous iron sucrose Administered at days 10 (±4) and 1 (±1) before the index procedure.
  Interventions: Drug: Erythropoietin
- Placebo (Placebo Comparator): Dosage: Saline solution 0.9% Administered at days 10 (±4) and 1 (±1) before the index procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erythropoietin — Combinaison drug of darboepoetin 0.75µg/Kg + 200mg intravenous iron sucrose
  Other Names: Darboepoetin
  Arms: Erythropoietin
Drug: Placebo — Saline solution 0.9%
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy of Erythropoietin (EPO) (+ iron) in reducing the rate of red blood cell transfusion requirements in patients with aortic stenosis undergoing transcatheter aortic valve replacement.

DETAILED DESCRIPTION:
STUDY DESIGN

Prospective randomized double blind study including patients diagnosed with severe symptomatic aortic stenosis and anemia undergoing aortic valve replacement. The patients will be identified in the cardiac surgery / aortic stenosis outpatient clinic or in the hospitalization department of the Institut Universitaire de Cardiologie et de Pneumologie de Quebec.

SAMPLE SIZE

100 patients (50 patients per group).

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥60-year old
2. Symptomatic aortic stenosis with a clinical indication for transcatheter aortic valve replacement, regardless of simultaneous percutaneous coronary intervention
3. Anemia defined according to the World Health Organization (WHO) definition 69:

   1. Men: Hemoglobin<130 g/L
   2. Women: <120 g/L

Exclusion Criteria:

1. Contraindication for transcatheter aortic valve replacement.
2. Erythropoietin treatment within last 30 days before Aortic Valve Replacement
3. Known anemia due to aplasia, other hemoglobinopathy or active bleeding requiring blood transfusion within last 30 days before Aortic Valve Replacement
4. Ferritin>800 µg/L
5. Uncontrolled hypertension (Blood pressure>175/95 )
6. Platelet count>450,000/L
7. Recent myocardial infarction requiring percutaneous coronary intervention or disabling stroke (within the last 30 days)
8. Dialysis patients
9. Hemodynamic instability as defined as the need of hemodynamic support with inotropic drugs, intraortic balloon pump counter-pulsation or left ventricular assist device before index procedure
10. Active cancer or very high risk of thromboembolic events
11. Known allergy or hypersensitivity to intravenous iron or Erythropoietin therapy
12. No written consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Rate of red blood cell transfusion | 30 days

SECONDARY OUTCOMES:
Number of packets of red cells | 30 days
Hemoglobin value | One day before index procedure
  Analysis g/L
Hemoglobin value | For the duration of hospital stay, an expected average of 1 week
Peak of troponin and creatinine kinase | For the duration of hospital stay, an expected average of 1 week
Incidence of acute kidney injury | At 48 hours following procedure
  Acute kidney injury defined as >25% decrease of estimated glomerular filtration rate (eGFR)
Need of hemodialysis | For the duration of hospital stay, an expected average of 1 week
Rate of new onset atrial fibrillation | For the duration of hospital stay, an expected average of 1 week
Days of hospital stay | For the duration of hospital stay, an expected average of 1 week
Days of intensive unit care stay | For the duration of hospital stay, an expected average of 1 week
Mortality | At 30-day, 1-year
Quality of life | At 30-day, 6-month, 1-year
  Questionnaire, Visual scale
Cost-effectiveness analysis of Erythropoietin-therapy | For the duration of hospital stay, an expected average of 1 week
Stroke rate | At 30-day

CONTACTS AND LOCATIONS:
Overall Officials: Josep Rodes Cabau, MD, Principal Investigator — Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Canada

REFERENCES:
- [Background] Karkouti K, Wijeysundera DN, Beattie WS; Reducing Bleeding in Cardiac Surgery (RBC) Investigators. Risk associated with preoperative anemia in cardiac surgery: a multicenter cohort study. Circulation. 2008 Jan 29;117(4):478-84. doi: 10.1161/CIRCULATIONAHA.107.718353. Epub 2008 Jan 2. PMID 18172032
- [Background] Kulier A, Levin J, Moser R, Rumpold-Seitlinger G, Tudor IC, Snyder-Ramos SA, Moehnle P, Mangano DT; Investigators of the Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. Impact of preoperative anemia on outcome in patients undergoing coronary artery bypass graft surgery. Circulation. 2007 Jul 31;116(5):471-9. doi: 10.1161/CIRCULATIONAHA.106.653501. Epub 2007 Jul 9. PMID 17620512
- [Background] Karkouti K, Djaiani G, Borger MA, Beattie WS, Fedorko L, Wijeysundera D, Ivanov J, Karski J. Low hematocrit during cardiopulmonary bypass is associated with increased risk of perioperative stroke in cardiac surgery. Ann Thorac Surg. 2005 Oct;80(4):1381-7. doi: 10.1016/j.athoracsur.2005.03.137. PMID 16181875
- [Background] Van Mieghem NM, Nuis RJ, Tzikas A, Piazza N, Schultz C, Serruys PW, de Jaegere PP. Prevalence and prognostic implications of baseline anaemia in patients undergoing transcatheter aortic valve implantation. EuroIntervention. 2011 Jun;7(2):184-91. doi: 10.4244/EIJV7I2A32. PMID 21646060
- [Background] van Straten AH, Hamad MA, van Zundert AJ, Martens EJ, Schonberger JP, de Wolf AM. Preoperative hemoglobin level as a predictor of survival after coronary artery bypass grafting: a comparison with the matched general population. Circulation. 2009 Jul 14;120(2):118-25. doi: 10.1161/CIRCULATIONAHA.109.854216. Epub 2009 Jun 29. PMID 19564556
- [Background] Society of Thoracic Surgeons Blood Conservation Guideline Task Force; Ferraris VA, Brown JR, Despotis GJ, Hammon JW, Reece TB, Saha SP, Song HK, Clough ER; Society of Cardiovascular Anesthesiologists Special Task Force on Blood Transfusion; Shore-Lesserson LJ, Goodnough LT, Mazer CD, Shander A, Stafford-Smith M, Waters J; International Consortium for Evidence Based Perfusion; Baker RA, Dickinson TA, FitzGerald DJ, Likosky DS, Shann KG. 2011 update to the Society of Thoracic Surgeons and the Society of Cardiovascular Anesthesiologists blood conservation clinical practice guidelines. Ann Thorac Surg. 2011 Mar;91(3):944-82. doi: 10.1016/j.athoracsur.2010.11.078. PMID 21353044
- [Background] Murphy GJ, Reeves BC, Rogers CA, Rizvi SI, Culliford L, Angelini GD. Increased mortality, postoperative morbidity, and cost after red blood cell transfusion in patients having cardiac surgery. Circulation. 2007 Nov 27;116(22):2544-52. doi: 10.1161/CIRCULATIONAHA.107.698977. Epub 2007 Nov 12. PMID 17998460
- [Background] Bucerius J, Gummert JF, Borger MA, Walther T, Doll N, Onnasch JF, Metz S, Falk V, Mohr FW. Stroke after cardiac surgery: a risk factor analysis of 16,184 consecutive adult patients. Ann Thorac Surg. 2003 Feb;75(2):472-8. doi: 10.1016/s0003-4975(02)04370-9. PMID 12607656
- [Background] Paone G, Brewer R, Theurer PF, Bell GF, Cogan CM, Prager RL; Michigan Society of Thoracic and Cardiovascular Surgeons. Preoperative predicted risk does not fully explain the association between red blood cell transfusion and mortality in coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2012 Jan;143(1):178-85. doi: 10.1016/j.jtcvs.2011.09.015. Epub 2011 Oct 19. PMID 22014719
- [Background] Koch CG, Li L, Van Wagoner DR, Duncan AI, Gillinov AM, Blackstone EH. Red cell transfusion is associated with an increased risk for postoperative atrial fibrillation. Ann Thorac Surg. 2006 Nov;82(5):1747-56. doi: 10.1016/j.athoracsur.2006.05.045. PMID 17062241
- [Background] Surgenor SD, DeFoe GR, Fillinger MP, Likosky DS, Groom RC, Clark C, Helm RE, Kramer RS, Leavitt BJ, Klemperer JD, Krumholz CF, Westbrook BM, Galatis DJ, Frumiento C, Ross CS, Olmstead EM, O'Connor GT. Intraoperative red blood cell transfusion during coronary artery bypass graft surgery increases the risk of postoperative low-output heart failure. Circulation. 2006 Jul 4;114(1 Suppl):I43-8. doi: 10.1161/CIRCULATIONAHA.105.001271. PMID 16820613
- [Background] Bagur R, Webb JG, Nietlispach F, Dumont E, De Larochelliere R, Doyle D, Masson JB, Gutierrez MJ, Clavel MA, Bertrand OF, Pibarot P, Rodes-Cabau J. Acute kidney injury following transcatheter aortic valve implantation: predictive factors, prognostic value, and comparison with surgical aortic valve replacement. Eur Heart J. 2010 Apr;31(7):865-74. doi: 10.1093/eurheartj/ehp552. Epub 2009 Dec 27. PMID 20037180
- [Background] Yoo YC, Shim JK, Kim JC, Jo YY, Lee JH, Kwak YL. Effect of single recombinant human erythropoietin injection on transfusion requirements in preoperatively anemic patients undergoing valvular heart surgery. Anesthesiology. 2011 Nov;115(5):929-37. doi: 10.1097/ALN.0b013e318232004b. PMID 22027622
- [Background] Kiyama H, Ohshima N, Imazeki T, Yamada T. Autologous blood donation with recombinant human erythropoietin in anemic patients. Ann Thorac Surg. 1999 Nov;68(5):1652-6. doi: 10.1016/s0003-4975(99)00755-9. PMID 10585037
- [Background] Sowade O, Warnke H, Scigalla P, Sowade B, Franke W, Messinger D, Gross J. Avoidance of allogeneic blood transfusions by treatment with epoetin beta (recombinant human erythropoietin) in patients undergoing open-heart surgery. Blood. 1997 Jan 15;89(2):411-8. PMID 9002942
- [Background] Gombotz H. Subcutaneous epoetin alfa as an adjunct to autologous blood donation before elective coronary artery bypass graft surgery. Semin Hematol. 1996 Apr;33(2 Suppl 2):69-70; discussion 71-2. PMID 8723587
- [Background] Weltert L, D'Alessandro S, Nardella S, Girola F, Bellisario A, Maselli D, De Paulis R. Preoperative very short-term, high-dose erythropoietin administration diminishes blood transfusion rate in off-pump coronary artery bypass: a randomized blind controlled study. J Thorac Cardiovasc Surg. 2010 Mar;139(3):621-6; discussion 626-7. doi: 10.1016/j.jtcvs.2009.10.012. Epub 2009 Dec 29. PMID 20042202
- [Background] Yazicioglu L, Eryilmaz S, Sirlak M, Inan MB, Aral A, Tasoz R, Eren NT, Kaya B, Akalin H. Recombinant human erythropoietin administration in cardiac surgery. J Thorac Cardiovasc Surg. 2001 Oct;122(4):741-5. doi: 10.1067/mtc.2001.115426. PMID 11581607
- [Background] Kyo S, Omoto R, Hirashima K, Eguchi S, Fujita T. Effect of human recombinant erythropoietin on reduction of homologous blood transfusion in open-heart surgery. A Japanese Multicenter study. Circulation. 1992 Nov;86(5 Suppl):II413-8. PMID 1424032
- [Derived] Nishiwaki H, Abe Y, Suzuki T, Hasegawa T, Levack WM, Noma H, Ota E. Erythropoiesis-stimulating agents for preventing acute kidney injury. Cochrane Database Syst Rev. 2024 Sep 20;9(9):CD014820. doi: 10.1002/14651858.CD014820.pub2. PMID 39301879